CLINICAL TRIAL: NCT02928614
Title: Biomarkers in Obese Patients With Knee Osteoarthritis Following Long-term Weight Maintenance
Brief Title: Biomarkers in Obese Patients With Knee Osteoarthritis; Weight Maintenance
Acronym: BIO-LOSEIT-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henrik Gudbergsen (Other)
Responsible Party: Sponsor-Investigator, Henrik Gudbergsen, MD, PhD, Parker Research Institute
Organization: Parker Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 137.08
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis; Obesity
Keywords: Osteoarthritis; Obesity; Liraglutide 3 mg; Liraglutide; Biomarkers
MeSH Terms: conditions — Osteoarthritis; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide 3 mg (Experimental): Arm description: Subjects will be up titrated to liraglutide 3 mg QD and stay on that dose for the remainder of the 52-week drug intervention period.
  Drug: Liraglutide 3 mg QD administered in a 6 mg/mL, 3 mL pen for subcutaneous injection.
  Dose escalation scheme: Initial dosage of 0.6 mg per day, escalated bi-weekly by 0.6 mg to 3 mg per day over a total of 8 weeks.
  Interventions: Drug: Liraglutide 3 mg (Saxenda)
- Liraglutide 3 mg placebo (Placebo Comparator): Arm description: Subjects will be up titrated to liraglutide 3 mg placebo QD and stay on that dose for the remainder of the 52-week drug intervention period.
  Drug: Liraglutide 3 mg placebo QD administered in a 6 mg/mL drug equivalent volumes, 3 mL pen for subcutaneous injection.
  Dose escalation scheme: Initial dosage of a 0.6 mg drug equivalent volume per day, escalated bi-weekly by an 0.6 mg drug equivalent volume per day to a 3 mg drug equivalent volume per day over a total of 8 weeks.
  Interventions: Drug: Liraglutide 3 mg placebo

INTERVENTIONS:
Drug: Liraglutide 3 mg (Saxenda)
  Arms: Liraglutide 3 mg
Drug: Liraglutide 3 mg placebo
  Arms: Liraglutide 3 mg placebo

SUMMARY:
This is a substudy to a randomized trial investigating the effect of liraglutide on body weight and pain in overweight or obese patients with knee osteoarthritis (NCT02905864). In the parent trial, patients will be subjected to an 8-week diet intervention phase including a low-calorie diet and dietetic counseling, after which they will be randomized to receive either liraglutide 3 mg or liraglutide 3 mg placebo as an add-on to dietetic guidance on re-introducing regular foods and a focus on continued motivation to engage in a healthy lifestyle.

This substudy aims to investigate the impact of, and subsequent change of biomarkers in obese patients with knee osteoarthritis following a randomization to Liraglutide 3 mg or Liraglutide 3 mg placebo treatment between weeks 0-52.

ELIGIBILITY:
Inclusion Criteria:

* Same as parent trial (NCT02905864)

Exclusion Criteria:

* Same as parent trial (NCT02905864)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in collagen II degradation fragment α-C2M | Week 0 to 52
  Blood sampling

SECONDARY OUTCOMES:
Change in collagen II degradation fragment β-C2M | Week 0 to 52
  Blood sampling
Change in non-coding RNA type snoRNAs U38 and U48 | Week 0 to 52
  Blood sampling
Change in miRNA-454 | Week 0 to 52
  Blood sampling
Change in miRNA let-7e | Week 0 to 52
  Blood sampling
Change in Nesfatin-1 | Week 0 to 52
  Blood sampling

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Frederiksberg, Capital Region, Denmark